CLINICAL TRIAL: NCT00467142
Title: Phase II Study Evaluating the Efficacy and Tolerance to Chemotherapy With 5-fluorouracil, Folinic Acid, Irinotecan and Bevacizumab as First-line Treatment in Patients With Metastatic Colorectal Cancer
Brief Title: Bevacizumab and Combination Chemotherapy as First-Line Therapy in Treating Patients With Metastatic Colorectal Cancer That Cannot Be Removed by Surgery
Acronym: OMEGA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000540522; IB-2006-31; IB-OMEGA; INCA-RECF0387; EUDRACT-2006-003901-22
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Results first posted 2022-04-20 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Fluorouracil; Irinotecan; Leucovorin; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Folfiri and Bevacizumab (Experimental): * Premedication = Dexchlorpheniramine, 5 mg in slow Direct IntraVeinous (DIV) on D1.
  * FOLFIRI (simplified LV5FU2 + irinotecan):
  * Irinotecan (Campto®): 180 mg/m² on D1 by IV infusion in 250 mL of 0.9% saline over 90 minutes.
  * LV5FU2, in its so-called "simplified" version, will be administered as follows L-folinic acid, as a 2-hour intravenous infusion, at a dose of 200 mg/m², on Day 1, in 500 mL of 5% glucose solution, concomitantly with the irinotecan infusion via a Y-tube, followed by 5 Fluorouracil (5 FU), intravenous bolus, at a dose of 400 mg/m² on D1, followed by 5 Fluorouracil (5 FU) as a 46-hour continuous infusion at a dose of 2400 mg/m² from D1 to D3, either in 1000 mL of 5% glucose solution, or in an electric syringe or pump dispenser
  * Bevacizumab (Avastin®): 5 mg/kg IV infusion in 100 mL of 0.9% saline over 90 minutes for the first infusion, then 60 minutes for the second infusion if tolerated, and 30 minutes for subsequent infusions if tolerated.
  Interventions: Biological: bevacizumab; Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Genetic: polymorphism analysis

INTERVENTIONS:
Biological: bevacizumab
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium
Genetic: polymorphism analysis

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of colorectal cancer by blocking blood flow to the tumor. Drugs used in chemotherapy, such as irinotecan, leucovorin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with combination chemotherapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving bevacizumab together with combination chemotherapy works as first-line therapy in treating patients with metastatic colorectal cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of bevacizumab, irinotecan hydrochloride, leucovorin calcium, and fluorouracil, in terms of partial or complete response, in patients with unresectable metastatic colorectal cancer.

Secondary

* Determine the duration of response in patients treated with this regimen.
* Determine the overall survival and progression-free survival of patients treated with this regimen.
* Determine the tolerability of this regimen in these patients.
* Assess the pharmacogenetics and change in genetic polymorphisms susceptible to modification by this regimen.

OUTLINE: This is a nonrandomized, multicenter study.

Patients receive irinotecan hydrochloride IV over 90 minutes, leucovorin calcium IV over 2 hours, and bevacizumab IV on day 1. Patients also receive fluorouracil IV over 46 hours beginning on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.

Blood and tissue samples are collected periodically for pharmacogenetic and genetic polymorphism analysis.

PROJECTED ACCRUAL: A total of 61 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon or rectum

  * No other histological types
* Metastatic, unresectable disease

  * No bone metastases only
* Unidimensionally measurable metastatic disease
* No CNS metastases

PATIENT CHARACTERISTICS:

* WHO performance status (PS) 0-2 OR Karnofsky PS 70-100%
* Life expectancy ≥ 12 weeks
* ANC > 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL
* Bilirubin ≤ 1.25 times normal (1.5 times normal in presence of hepatic metastases)
* AST and ALT < 3 times normal (5 times normal in presence of hepatic metastases)
* Creatinine < 1.25 times normal
* No proteinuria
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other cancer in the past 5 years except for carcinoma in situ of the uterine cervix or basal cell skin cancer
* No hypersensitivity to fluorouracil
* No hypersensitivity to leucovorin calcium, bevacizumab, or their excipients
* No hypersensitivity to Chinese hamster ovarian cell products or other recombinant humanized or nonhumanized monoclonal antibodies
* No allergy to irinotecan hydrochloride
* No prior reaction to attenuated vaccines (fever, jaundice)
* No poor nutritional status
* No Biermer anemia or other anemia due to vitamin B12 deficiency
* No uncontrolled symptomatic occlusion or subocclusion
* No medullary hypoplasia or severe insufficiency
* No prior chronic intestinal disease
* No Gilbert's syndrome
* No intra-abdominal inflammatory reaction (e.g., gastroduodenal ulcer, diverticulitis, or colitis)
* No chronic intestinal inflammatory disease
* No thromboembolic arterial condition in the past 6 months, including any of the following:

  * Cardiovascular accident
  * Transient ischemic attack
  * Myocardial infarction
* No infection or serious noncancerous disease
* No condition that is unstable or would increase risk to the patient, including any of the following:

  * Unstable angina
  * Poorly controlled hypertension
  * Severe cardiac insufficiency
  * Serious arrhythmia
  * Bleeding diathesis
  * Pulmonary disease at risk of decompensation
* No familial, geographical, social, or psychological condition that would preclude study participation
* No prisoners or patients without guardians

PRIOR CONCURRENT THERAPY:

* At least 8 weeks since prior surgery
* At least 6 months since prior adjuvant chemotherapy
* At least 1 month since prior palliative chemotherapy
* No prior abdominal or pelvic radiotherapy
* At least 30 days since prior participation in another investigational study
* No prior bevacizumab
* No extensive intestinal resection (e.g., partial colectomy or extensive thin resection)
* No concurrent warfarin, Hypericum perforatum (St. John's wort), or prophylactic phenytoin

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-01-23 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yves Becouarn, MD, Study Chair — Institut Bergonié
Locations (1):
- Institut Bergonie, Bordeaux, France

REFERENCES:
- [Result] Becouarn Y, Cany L, Pulido M, Beyssac R, Texereau P, Le Morvan V, Bechade D, Brunet R, Aitouferoukh S, Lalet C, Mathoulin-Pelissier S, Fonck M, Robert J. FOLFIRI(R) and bevacizumab in first-line treatment for colorectal cancer patients: safety, efficacy and genetic polymorphisms. BMC Res Notes. 2014 Apr 23;7:260. doi: 10.1186/1756-0500-7-260. PMID 24758527

RESULTS

PARTICIPANT FLOW:
Groups:
- Folfiri and Bevacizumab: * Premedication = Dexchlorpheniramine, 5 mg in slow Direct IntraVeinous (DIV) on D1.
  * FOLFIRI (simplified LV5FU2 + irinotecan):
  * Irinotecan (Campto®): 180 mg/m² on D1 by IV infusion in 250 mL of 0.9% saline over 90 minutes.
  * LV5FU2, in its so-called "simplified" version, will be administered as follows L-folinic acid, as a 2-hour intravenous infusion, at a dose of 200 mg/m², on Day 1, in 500 mL of 5% glucose solution, concomitantly with the irinotecan infusion via a Y-tube, followed by 5 Fluorouracil (5 FU), intravenous bolus, at a dose of 400 mg/m² on D1, followed by 5 Fluorouracil (5 FU) as a 46-hour continuous infusion at a dose of 2400 mg/m² from D1 to D3, either in 1000 mL of 5% glucose solution, or in an electric syringe or pump dispenser
  * Bevacizumab (Avastin®): 5 mg/kg IV infusion in 100 mL of 0.9% saline over 90 minutes for the first infusion, then 60 minutes for the second infusion if tolerated, and 30 minutes for subsequent infusions if tolerated.
  bevacizumab
  fluorouracil
  irinotecan hydrochloride
  leucovorin calcium
  polymorphism analysis
Period: Overall Study
Arm/Group | Folfiri and Bevacizumab
Started | 62
Completed | 59
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Folfiri and Bevacizumab
Number analyzed (Participants) | 62
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67.9 [60.4 to 75.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 25
Region of Enrollment [Number; unit: participants]
  France | 62

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Objective Response (Partial or Complete Responses)
Description: Objective response defined as complete or partial responses according to RECIST v1.0. Complete response is defined as the disappearance of all target lesions and partial response is defined as at least a 30% decrease in the sum of the longest diameters (SLD) of target lesions, taking as reference the baseline SLD (RECIST V1.0.).Radiologic assessment was carried out every four cycles (8 weeks) with centralized external secondary review.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Folfiri and Bevacizumab
Number analyzed (Participants) | 59
percentage of participants | 47.5 [34.3 to 60.9]

2. Secondary Outcome: Median Duration of Response
Description: Duration of response is defined as the delay between response (complete or partial) and disease progression according to RECIST V1.0. Therefore, this criterion can only be assessed in in subjects who have responded. Complete response is defined as the disappearance of all target lesions and partial response is defined as at least a 30% decrease in the sum of the longest diameters (SLD) of target lesions, taking as reference the baseline SLD (RECIST V1.0.). Progression is defined as a 20% increase in the sum of the longest diameters (SLD) of target lesions, taking as reference the baseline SLD, or appearance of one or several new lesions (RECIST V1.0) Radiologic assessment was carried out every four cycles (8 weeks) with centralized external secondary review.
Time Frame: 24 months
Population: 28 patients in partial response were evaluable for median duration of response.
Measure: Median (Full Range); unit: months
Arm/Group | Folfiri and Bevacizumab
Number analyzed (Participants) | 28
months | 9.5 [2.7 to 20]

ADVERSE EVENTS:
Description: Only serious adverse events were monitored. Adverse events (non-serious) were not assessed/monitored during the study.
Arm/Group | Folfiri and Bevacizumab
Serious Adverse Events (participants affected / at risk) | 20/62
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Folfiri and Bevacizumab (N=62)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Colitis (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Obstruction (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Bronchial infection (Infections and infestations) | 2 (3)
Phlebitis (Vascular disorders) | 2 (2)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Breast infection (Infections and infestations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
RESTORATION OF COLORECTAL CONTINUITY (Injury, poisoning and procedural complications) | 1 (1)
PORTAL EMBOLISATION (Injury, poisoning and procedural complications) | 1 (1)
White blood cell decreased (Blood and lymphatic system disorders) | 1 (1)
DETERIORATION OF GENERAL HEALTH STATUS (General disorders) | 1 (1)
Atrial fibrillaton (Cardiac disorders) | 1 (1)
Myocardial infarction (Vascular disorders) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes